CLINICAL TRIAL: NCT02003833
Title: Randomized, Controlled, Multi-Centered, Double-Blind Investigation of Injectable Poly-L-Lactic Acid (Sculptra Aesthetic) for Improving Facial Wrinkles and Skin Quality
Brief Title: Poly-L-lactic Acid for Skin Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sadick Research Group (Other)
Responsible Party: Principal Investigator, Neil Sadick, Medical Director, Sadick Research Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLLA SkinQ
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Skin Aging
Keywords: Poly-L-lactic acid; Sculptra Aesthetic; Skin Quality; Wrinkles; Filler

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Poly-L-lactic acid (Experimental): Subjects in the treatment arm will receive three injections of 5 cc of poly-L-lactic acid (PLLA) into both sides of the face.
  Interventions: Device: Poly-L-lactic acid
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive three injections of 5 cc of saline into both sides of the face. After the completion of the study, subjects in the placebo arm will receive free injections with Sculptra Aesthetic same as the treatment arm.
  Interventions: Device: Placebo comparator

INTERVENTIONS:
Device: Poly-L-lactic acid — Sculptra injections
  Other Names: Sculptra Aesthetic; P030050/S002
  Arms: Poly-L-lactic acid
Device: Placebo comparator — saline injections
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Anecdotal evidence suggests that patients' skin quality may improve as a result of poly-L-lactic acid injection. While this is not the primary goal of such treatments it is often seen and described as so called "Sculptra glow".

The aim of this study is to evaluate the effect of repeated subcutaneous injections of poly-L-lactic acid (Sculptra Aesthetic) on skin quality.

Participating subjects will be part of the study for about 15 months. There will be an initial treatment period of up to 12 weeks, followed by a 12-month follow-up period. There will be a total of 7 scheduled visits.

This study is a double-blind, randomized study. "Double-blind" means that neither the subjects nor the study doctor will know who is receiving Sculptra Aesthetic or placebo. "Randomized" means that the group subjects will be placed in is decided by chance, similar to drawing numbers out of a hat or flipping a coin. Subjects will have a 1 out of 2 chance of receiving the active study drug. After the completion of the study, if subjects are assigned to the control (placebo) group they will receive free injections with Sculptra Aesthetic same as the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization
* Healthy females between 30 and 60 years of age
* Subjects with Fitzpatrick photo skin types I-IV
* Subjects with shallow to deep nasolabial fold contour deficiencies or other facial wrinkles
* Subjects who agree not to have any procedures affecting facial wrinkles (e.g. filler, botulinum toxin, radiofrequency, laser, IPL, ultrasound) for the duration of the study
* Subjects who do agree not to have any other procedures affecting skin quality (microdermabrasion, peels, acne treatments, etc.) for the duration of the study
* Subjects who understand this study and are able to follow study instructions and are willing to attend the required study visits
* Subjects who agree to be photographed for research reasons and their identity may not be concealed in these photographs.

Exclusion Criteria:

* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
* Subjects who cannot understand or are not willing to comply with the requirements of the study
* Subjects who have a known allergy to poly-L-lactic acid, carboxymethylcellulose, non-pyrogenic mannitol or any anesthetic
* Subjects who have taken any NSAIDs (aspirin, ibuprofen, etc.) within 7 days before treatment
* Subjects who have taken acetaminophen 24 hours before treatment
* Subjects who have had fillers or botulinum toxin in the treatment area in the past 12 months
* Subjects who have had treatments with poly-L-lactic acid in the face at any time
* Subjects who have had any kind of facial dermabrasion, chemical peel, laser, or IPL treatment including superficial treatments for aesthetic reasons in the past 6 months or for the duration of the study
* Subjects who does not agree to avoid using tanning beds or intensive exposure to the sun 2 two weeks prior to each office visit.
* Subjects who have any dermatologic conditions including acne, rosacea, eczema, psoriasis, actinic keratosis, severe sun damage, infection or scars within the treatment area
* Subjects who have an active inflammatory process (skin eruptions such as cysts, pimples, rashes or hives) or infection within the treatment area
* Subjects who have any known cancer including skin cancers (basal cell carcinoma, squamous cell carcinoma and melanoma)
* Subjects who have had systemic corticosteroid therapy in the past 6 months or for the duration of the study
* Subjects with a known history of poor wound healing
* Subjects with a known history of keloids (excessive scarring)
* Subjects who are HIV positive
* Subjects who have an existing medical condition that the Investigator considers may put the subject at risk or compromise their participation in the study
* Subjects who have participated in another research study in the past 30 days
* Subjects who are currently involved in any injury litigation claims

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement in skin quality | 15 months
  The primary endpoint is defined as the degree of improvement in skin quality measured by a blinded, trained evaluator using standardized pictures as well as live evaluations rated by a blinded investigator and the subjects

SECONDARY OUTCOMES:
Improvement of skin physiology | 15 months
  Non-invasive biophysical measurements will be used to assess sub-clinical changes in skin quality including skin hydration, elasticity, density and dermal thickness and a decrease in transepidermal water loss
Investigator and patient satisfaction | 15 months
  Investigator and patient satisfaction will be assessed with a quartile scale.
Safety of repeated injections with Sculptra Aesthetic | 15 months
  Safety analyses will be done on all treated patients, defined by any subject who received at least one study treatment. Compiled side effects, including all expected or unexpected side effects but not limited to site discomfort, redness, bruising, bleeding, itching, and swelling, small and larger lumps under the skin

CONTACTS AND LOCATIONS:
Overall Officials: Neil S Sadick, MD, Principal Investigator — Sadick Research Group; William Hanke, MD, Principal Investigator — Laser and Skin Surgery Center of Indiana
Locations (2):
- United States (2):
  - Laser and Skin Surgery Center of Indiana, Carmel, Indiana
  - Sadick Research Group, New York, New York

REFERENCES:
- See also: Laser and Skin Surgery Center of Indiana — http://www.thelassi.com/